CLINICAL TRIAL: NCT00007410
Title: Genetic Architecture of Plasma T-PA and PAI-1
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 959; R01HL065234 (NIH)
Record Dates: First submitted 2000-12-19; First posted 2000-12-19 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Thrombosis; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Thrombosis; Atherosclerosis

SUMMARY:
To determine the effects of six genes on thrombotic risk factors known to be associated with the development of heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

Abnormalities in the plasminogen activator system have been implicated in the pathogenesis of arterial and cerebral thrombosis. In particular, elevated plasma levels of plasminogen activator inhibitor-1 (PAI-1), tissue-type plasminogen activator (t-PA), and t-PA/PAI-1 complexes have been found to correlate with increased risk of myocardial infarction (MI) and/or stroke. Vascular fibrinolytic balance is, to a large part, determined by the competing effects of t-PA and PAI-1, and reflects a complex interplay between genetic and environmental factors. The present collaboration focuses on the common hypothesis that the association between activation of the renin-angiotensin-aldosterone system (RAAS) and atherothrombotic events derives from an interaction between the RAAS and the fibrinolytic system.

The study is part of an initiative "Thrombosis of the Arterial and Cerebral Vasculature: New Molecular Genetic Concepts for Prevention and Treatment" which was released in April 1999. The objective of the initiative is to establish collaborative teams of closely interacting investigators with diverse, complementary areas of expertise to elucidate the molecular genetic mechanisms of thrombosis in the arterial and cerebral vasculature.

DESIGN NARRATIVE:

The investigators will use two population-based samples of unrelated individuals to address their aims: 1) study subjects in the PREVEND study in Groningen, The Netherlands in whom DNA and plasma samples and clinical data have already been collected and 2) an estimated 2000 unrelated study subjects from Ghana, Africa in whom data need to be collected. The collaborative study focuses on the common hypothesis that the association between activation of the renin-angiotensin-aldosterone system (RAAS) and atherothrombotic events derives from an interaction between the RAAS and the fibrinolytic system.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Moore — Vanderbilt University

REFERENCES:
- [Background] Moore JH, Williams SM. New strategies for identifying gene-gene interactions in hypertension. Ann Med. 2002;34(2):88-95. doi: 10.1080/07853890252953473. PMID 12108579
- [Background] Hahn LW, Ritchie MD, Moore JH. Multifactor dimensionality reduction software for detecting gene-gene and gene-environment interactions. Bioinformatics. 2003 Feb 12;19(3):376-82. doi: 10.1093/bioinformatics/btf869. PMID 12584123
- [Background] Ritchie MD, Hahn LW, Moore JH. Power of multifactor dimensionality reduction for detecting gene-gene interactions in the presence of genotyping error, missing data, phenocopy, and genetic heterogeneity. Genet Epidemiol. 2003 Feb;24(2):150-7. doi: 10.1002/gepi.10218. PMID 12548676
- [Background] Moore JH, Smolkin ME, Lamb JM, Brown NJ, Vaughan DE. The relationship between plasma t-PA and PAI-1 levels is dependent on epistatic effects of the ACE I/D and PAI-1 4G/5G polymorphisms. Clin Genet. 2002 Jul;62(1):53-9. doi: 10.1034/j.1399-0004.2002.620107.x. PMID 12123488
- [Background] Coffey CS, Hebert PR, Krumholz HM, Morgan TM, Williams SM, Moore JH. Reporting of model validation procedures in human studies of genetic interactions. Nutrition. 2004 Jan;20(1):69-73. doi: 10.1016/j.nut.2003.09.012. No abstract available. PMID 14698017
- [Background] Moore JH, Hahn LW. Petri net modeling of high-order genetic systems using grammatical evolution. Biosystems. 2003 Nov;72(1-2):177-86. doi: 10.1016/s0303-2647(03)00142-4. PMID 14642666
- [Background] Moore JH. The ubiquitous nature of epistasis in determining susceptibility to common human diseases. Hum Hered. 2003;56(1-3):73-82. doi: 10.1159/000073735. PMID 14614241
- [Background] Ritchie MD, White BC, Parker JS, Hahn LW, Moore JH. Optimization of neural network architecture using genetic programming improves detection and modeling of gene-gene interactions in studies of human diseases. BMC Bioinformatics. 2003 Jul 7;4:28. doi: 10.1186/1471-2105-4-28. Epub 2003 Jul 7. PMID 12846935
- [Background] Williams SM, Ritchie MD, Phillips JA 3rd, Dawson E, Prince M, Dzhura E, Willis A, Semenya A, Summar M, White BC, Addy JH, Kpodonu J, Wong LJ, Felder RA, Jose PA, Moore JH. Multilocus analysis of hypertension: a hierarchical approach. Hum Hered. 2004;57(1):28-38. doi: 10.1159/000077387. PMID 15133310
- [Background] Smith MW, Patterson N, Lautenberger JA, Truelove AL, McDonald GJ, Waliszewska A, Kessing BD, Malasky MJ, Scafe C, Le E, De Jager PL, Mignault AA, Yi Z, De The G, Essex M, Sankale JL, Moore JH, Poku K, Phair JP, Goedert JJ, Vlahov D, Williams SM, Tishkoff SA, Winkler CA, De La Vega FM, Woodage T, Sninsky JJ, Hafler DA, Altshuler D, Gilbert DA, O'Brien SJ, Reich D. A high-density admixture map for disease gene discovery in african americans. Am J Hum Genet. 2004 May;74(5):1001-13. doi: 10.1086/420856. Epub 2004 Apr 14. PMID 15088270
- [Background] Moore JH, Ritchie MD. STUDENTJAMA. The challenges of whole-genome approaches to common diseases. JAMA. 2004 Apr 7;291(13):1642-3. doi: 10.1001/jama.291.13.1642. No abstract available. PMID 15069055
- [Background] Tsai CT, Lai LP, Lin JL, Chiang FT, Hwang JJ, Ritchie MD, Moore JH, Hsu KL, Tseng CD, Liau CS, Tseng YZ. Renin-angiotensin system gene polymorphisms and atrial fibrillation. Circulation. 2004 Apr 6;109(13):1640-6. doi: 10.1161/01.CIR.0000124487.36586.26. Epub 2004 Mar 15. PMID 15023884
- [Background] Zeng C, Sanada H, Watanabe H, Eisner GM, Felder RA, Jose PA. Functional genomics of the dopaminergic system in hypertension. Physiol Genomics. 2004 Nov 17;19(3):233-46. doi: 10.1152/physiolgenomics.00127.2004. PMID 15548830
- [Background] Moore JH. Computational analysis of gene-gene interactions using multifactor dimensionality reduction. Expert Rev Mol Diagn. 2004 Nov;4(6):795-803. doi: 10.1586/14737159.4.6.795. PMID 15525222
- [Background] Thornton-Wells TA, Moore JH, Haines JL. Genetics, statistics and human disease: analytical retooling for complexity. Trends Genet. 2004 Dec;20(12):640-7. doi: 10.1016/j.tig.2004.09.007. PMID 15522460
- [Background] Robinson M, Williams SM. Role of two angiotensinogen polymorphisms in blood pressure variation. J Hum Hypertens. 2004 Dec;18(12):865-9. doi: 10.1038/sj.jhh.1001768. PMID 15343353
- [Background] Hahn LW, Moore JH. Ideal discrimination of discrete clinical endpoints using multilocus genotypes. In Silico Biol. 2004;4(2):183-94. PMID 15107022
- [Background] Moore JH, Boczko EM, Summar ML. Connecting the dots between genes, biochemistry, and disease susceptibility: systems biology modeling in human genetics. Mol Genet Metab. 2005 Feb;84(2):104-11. doi: 10.1016/j.ymgme.2004.10.006. Epub 2004 Dec 19. PMID 15670716